CLINICAL TRIAL: NCT00451724
Title: Intranasal Ketamine for Procedural Sedation in Pediatric Laceration Repair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0014-07
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Laceration
Keywords: Prospective; Randomized; Double blinded; Sedation; Ketamine; Intranasal
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Intranasal ketamine

SUMMARY:
The purpose of this study is to compare how well three different doses of ketamine, given as a spray into the nose, help to sedate children and help them tolerate repairs of cuts on their faces.

DETAILED DESCRIPTION:
Procedural sedation is frequently used to facilitate distressing and painful procedures in the pediatric emergency department. However, administering an intramuscular medication or placing an intravenous line to give intravenous medications can be as distressing as the procedure itself. Oral medications generally take longer to work and are subject to first-pass metabolism. Another alternative is to give the medication by the intranasal route, which only requires a spray into the nose. Ketamine is a good sedative drug with favorable qualities, and is often used intramuscularly or intravenously. It has been used intranasally as a pre-induction by anesthetics, sedation for CT scans, and brief dental procedures, but its use has not yet been demonstrated in the setting of the pediatric emergency department for procedural sedation. We will be comparing three different doses of ketamine, applied intranasally using a mucosal atomization device, and determining if there are any differences in efficacy of sedation, time to onset of sedation, duration of sedation, caregiver and physician satisfaction, and number of adverse events. We will also use this opportunity to determine ketamine bioavailability when given intranasally using the mucosal atomization device.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 to 7 years old
* Simple facial laceration, defined as: linear; requiring two or more sutures; no greater than 5.0 centimeters; does not cross the lid margin of the eye; does not require a plastics/face surgery consult; occured within the last 24 hours.
* Physician feels that intravenous sedation is required to perform the laceration repair

Exclusion Criteria:

* Closed head injury, any alteration in level of consciousness, clinical suspicion of intracranial injury or increased intracranial pressure
* Any conditions that qualify patient as American Society of Anesthesiologists' (ASA) III or IV
* Known diagnoses of hyperthyroidism or porphyria
* Glaucoma or penetrating eye injury
* Hypertension
* Any contraindication, including drug allergy, to study medications
* Severe trauma with other injuries requiring operative intervention
* Abnormal neurological exam in a previously normal child

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2007-05; Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of sedation (OSBDR) | 30 minutes
Time to onset of sedation (Ramsay 6-point Sedation Scale) | 30 minutes

SECONDARY OUTCOMES:
Duration of sedation | Up to 1 hour
Primary caregiver satisfaction | 24 hours
Physician satisfaction | Duration of procedure
Ketamine bioavailability | 1 hour
Abnormalities in cardiopulmonary function | Until time of discharge
Administration of supplemental sedative medication | During time required for procedure
Prolonged sedation (i.e. > 1 hour) | Until time of discharge from emergency department

CONTACTS AND LOCATIONS:
Overall Officials: James G Linakis, PhD, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Hasbro Children's Hospital, Providence, Rhode Island, United States